CLINICAL TRIAL: NCT00462111
Title: Effect of Indomethacin on Reaction Time, Postural Balance and the Ability to Avoid Suddenly Appearing Obstacles During Gait in Healthy Middle-aged Individuals.
Brief Title: Indomethacin and Mechanisms Underlying Risk of Falling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: SKM002
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Healthy
Keywords: indometacin; reaction time; postural balance; obstacle avoidance; accidental falls
MeSH Terms: interventions — Indomethacin

INTERVENTIONS:
Drug: Indometacin

SUMMARY:
The purpose of this study is to determine whether indometacin has an effect on reaction time, postural stability, and the avoidance of obstacles.

DETAILED DESCRIPTION:
A lot of (epidemiologic) research is done on causes for falls and factors contributing to falling. Most of this research was conducted on the elderly, either community-dwelling or institutionalised. It became clear that the elderly have a greater risk at falling because of:

* physiological changes due to increasing age [Gerdhem et al., 2005]
* previous falls [Myers et al., 1991; Lipsitz et al., 1992]
* comorbidity (including RA) [Bergland et al., 2004; Gerdhem et al., 2005; Lawlor et al., 2003]
* polypharmacy [Lawlor et al., 2003; Walker et al., 2005; Ziere et al., 2005] and/or
* use of specific drugs like antidepressives, benzodiazepines, vasodilators, and NSAIDs [Cumming R, 1998; Herings RMC, 2001; Kallin K et al., 2004; Granek et al., 1987].

The relation between benzodiazepines and falling has been extensively investigated in and affirmed by several fields of research and is practically common sense. However, the (possible) relation between NSAIDs and falling is much less investigated, even though there are various articles in which a higher risk of falling when using NSAIDs is stated; sometimes the risk is even as high as with benzodiazepines [Cumming R, 1998; Granek et al., 1987; Walker et al., 2005].

Objective of the study:

NSAIDs are drugs that are often prescribed to patients with rheumatic or orthopedic diseases. They seem to be at a greater risk for falls than healthy persons because of their disease, age and medication use. Therefore it is very important to keep this risk as small as possible. In this study healthy adults are measured on reaction time, postural balance and obstacle avoidance with and without use of indometacin or placebo. This is done in order to gain more comprehension in the mechanism and actual risk for falls when using NSAIDs.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50-70 years old
* Not using any non-steroidal anti-inflammatory drugs (NSAIDs) for at least 3 days prior to the test session

Exclusion Criteria:

* Neurological or orthopedic disorders
* Poor comprehension of Dutch language
* Hearing problems
* Severe problems with heart and/or blood vessels
* Acutely existing ulcus ventriculi and/or duodeni, or history of ulcus
* Allergy against indomethacin, aspirin, or other NSAIDs
* Patients with nasal polyps reacting with an angioedema to other NSAIDs
* Severe preexisting renal and liver damage
* Co-medication
* Over 100 kg of weight

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Success rate on the obstacle avoidance task

SECONDARY OUTCOMES:
Reaction time
Root mean square (RMS) of the velocity and amplitude of the centre of pressure (COP)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques van Limbeek, MD, Principal Investigator — Sint Maartenskliniek; Jaak Duysens, Prof, Study Chair — St Maartenskliniek and University Medical Centre St. Radboud, Nijmegen
Locations (1):
- Sint Maartenskliniek, Nijmegen, Netherlands